CLINICAL TRIAL: NCT04180891
Title: Profiles of Empathy and Emotional Intelligence Promoted by Written Examination Combined to Oral Interviews During the Selection of 1st Year Health Students at the Paris University of Medicine
Brief Title: Empathy and Emotional Intelligence Promoted by the Selection Process in 1st Year of Health Studies at the Paris University Medical School
Acronym: PREMIS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Paris 5 - Rene Descartes (Other)
Responsible Party: Principal Investigator, Eloi Choisnet, resident, University of Paris 5 - Rene Descartes
Other Study IDs: Empathy 7
Record Dates: First submitted 2019-11-23; First posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Health Studies First-year Course Selection
Keywords: empathy; emotional intelligence; multiple mini-interviews

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- successful test: Students that have successfully passed the test procedure (directly with written exam or after written and oral interviews) and that can enter one of the four medical courses of health studies (medicine, pharmacy, dentistry, midwifery).
- failed test: Students that have failed to enter one of the four medical courses of health studies (medicine, pharmacy, dentistry, midwifery) after the selection procedure.

SUMMARY:
As the interpersonal skills such as empathy and emotional intelligence take more and more importance in the medical education, the Paris University of Medicine has introduced for the first time in 2019 some multiple mini-interviews (MMI) in addition to the traditional written examination, to graduate the 1st year student in health studies.

The selection process aims at promoting students with high academic results but also with good interpersonal abilities. In this new selection process, MMI will be used in addition to written tests, but only to attribute the last places available after a first ranking based on academic results.

So after the written examination, students with the best written exam marks will directly graduate, others will require MMI to graduate and some will directly fail.

The main hypothesis is that this selection procedure may promote stronger interpersonal abilities profiles in the group that succeed to enter one of the health studies course than in the group that failed.

This study will measure the clinical empathy and emotional intelligence abilities of all the 1st year students applying for this new selection process, using validate self-administered questionnaires.

Then the investigators will compare the scores of empathy and emotional intelligence in the group that succeed the selection process, to the group that failed. Furthermore, in the success group, the investigators will compare the scores between students that directly graduated and students that required MMI. Scores will also be compared considering some sociodemographic data.

The result of that studies could give strong arguments to modify the selection process and extend the use of MMI in medical school in France.

DETAILED DESCRIPTION:
INTRODUCTION : Considering empathy and emotional intelligence in the early stages of health studies has become a significant concern, all the more as empathy level among medicine students seems to decrease by the years. This loss of clinical empathy takes particularly place after the 3rd year of medicine studies, when students start being in contact with real patients. Starting from that, the investigators will study if the selection that occurs by the end of the 1st year of health studies in France, and which select students that can enter one of the course (medicine, dentistry, pharmacy, midwifery), is designed to promote not only academic skills but also interpersonal abilities. That selection procedure is especially important because it will determine the profiles of health professionals that will enter medical course and will be the future practitioner. In order to to consider more the interpersonal abilities of the students during the selection process, some Multiple Mini-Interview (MMI) have been introduced. The MMI will be used to attribute the last 20% of the places available (80% of the places will be directly attributed by the classic written examen)

METHODS : In this research, it will be proposed to all the 1st year health students registered in Paris University of medicine for the year 2019/2020 (about 1200 students) to complete four self-administered questionnaire : the Jefferson Scale of Empathy (student version),the Interpersonal Reactivity Index (IRI), the Questionnaire of Cognitive and Affective Empathy (QCAE) and the Emotional Expressivity Scale (EES). The students will get a personal access to the questionnaires by their digital workspace on the University's website. By the end of the year, they will be separated in 2 groups : students that have succeeded to the selection process and that can enter one of the health course, and students that failed. Then the investigators will compare the scores of the several self-administered questionnaires in the 2 groups.

OBJECTIVE : That study wants to determine if the selection process in first year of health student in the Paris University of Medicine is able to promote students profiles with strong interpersonal abilities so as academics skills. That study will also try to determine if the introduction of MMI has an impact on the empathy scores of the selected students.

ELIGIBILITY:
Inclusion Criteria:

* students registered in the first year of heath studies in Paris University Medical School

Exclusion Criteria:

* refusal of consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will come from the all students enrolled in first year of health studies in the Paris University of Medicine for the academic year 2019/2020.
  All of the students can enter the study if the answer the questionnaires, regardless of age or gender.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Empathy score | through study completion, an average of 1 year
  Empathy score will be measured by Jefferson Scale of Physician Empathy (JSPE) Student version and compared between group "success" and group "failure".

SECONDARY OUTCOMES:
Secondary empathy score (1) | through study completion, an average of 1 year
  Score at the Interpersonal Reactivity Index (IRI) compared between group "success" and group "failure".
Secondary empathy score (2) | through study completion, an average of 1 year
  Score at the Questionnaire of Cognitive and Affective Empathy (QCAE) compared between group "success" and group "failure".
Emotional intelligence score | through study completion, an average of 1 year
  Score at the Emotional Expressivity Scale (EES) compared between group "success" and group "failure".

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Jaury, Pr, Study Director — Paris Descartes University of Medicine
Locations (1):
- Paris University of Medicine, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No